CLINICAL TRIAL: NCT06826729
Title: The Characteristics of Blood Glucose Profile and the Changes of Endogenous and Exogenous Hormones in Patients with Post-chronic Pancreatitis Diabetes Mellitus
Brief Title: The Characteristics of Blood Glucose Profile and the Changes of Hormones in PPDM-C Population
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Tuo Li, MD, Prof., Shanghai Changzheng Hospital
Other Study IDs: 2024SL140
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-11

CONDITIONS: Chronic Pancreatitis; Diabetes
Keywords: chronic pancreatitis; PPDM-C; CGM
MeSH Terms: conditions — Pancreatitis, Chronic; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, urine and feces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study was to explore the characteristics of blood glucose spectrum, changes of endocrine/exocrine pancreatic function and the correlation between them in patients with PPDM-C.

DETAILED DESCRIPTION:
The benefits of this study to participants include:

1. It will help to make early diagnosis or risk screening for the potential related risks and concomitant diseases of the disease;
2. Provide necessary suggestions for the treatment and intervention of the disease, or provide useful information for the related research of the disease.
3. We will provide Abbott version h dynamic glucose meter and assessment of internal and external secretion function. The researcher will provide professional endocrine related lifestyle and drug guidance for the subjects according to their CGMS data.

The risks that this study may bring to participants are:

There may be some very small risks in specimen collection, including transient pain, local cyanosis, etc. a few people will have mild dizziness or extremely rare needle infection.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Chinese subjects;

  * Was ≥ 18 years old when signing the informed consent;

    * Patients with complete diagnosis of chronic pancreatitis; ④ Those who voluntarily signed informed consent; ⑤ Those who complete serum samples in multiple centers and put them into storage.

Exclusion Criteria:

* Patients with impaired glucose tolerance but undiagnosed diabetes;

  * Patients with T1DM related autoimmune markers or other types of DM;

    * Patients with autoimmune pancreatitis, recurrent acute pancreatitis or acute onset of chronic pancreatitis;

      * Patients who underwent pancreatic surgery or related invasive procedures during treatment;

        * Previous or current malignant tumor; ⑥ Pregnancy or lactation; ⑦ Suffering from severe heart, liver or kidney dysfunction or malignant disease; ⑧ Failure to sign informed consent for cognitive impairment or other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with chronic pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-02-11 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Blood glucose profile characteristics of patients with PPDM-C | From February 2025 to December 2025